CLINICAL TRIAL: NCT01050231
Title: Robotics For Rehabilitation Therapy: Functional Versus Individual Joint Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, David Reinkensmeyer, Professor of Mechanical and Aerospace Engineering, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HS#2005-4506
Record Dates: First submitted 2008-02-21; First posted 2010-01-15 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Cerebrovascular Accident
Keywords: stroke; cerebrovascular accident; robot
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic group (Type I) (Experimental): Type I Robotic Therapy (Functional activities first) Participants in this group will participate in functional/task-oriented multi-joint training with the BONES robot first, followed by individual joint training with the BONES robot. A one-week break was provided between interventions.
  Interventions: Device: Functional/ Multi-joints activities; Device: Individual Joint Training
- Robotic group (Type II) (Active Comparator): Type II Robotic Therapy (Individual joints first) Participants in this group will participate in individual joint training with the BONES robot first, followed by functional/task-oriented multi-joint training with the BONES robot. A one-week break was provided between interventions.
  Interventions: Device: Functional/ Multi-joints activities; Device: Individual Joint Training

INTERVENTIONS:
Device: Functional/ Multi-joints activities — Subjects participated in 4 weeks of robotic training with the device: BONES (Biomimetic Orthosis Neurorehabilitation for Elbow and Shoulder), 3 days per week, 1 hour per day with the robotic exercise program focusing on functional tasks such as cleaning the windows, driving a steering wheel, grocery shopping, etc.
Device: Individual Joint Training — Subjects participated in 4 weeks of training with the robotic device BONES, 3 days per week, 1 hour per day with a robot-assisted exercise program. The robotic exoskeleton assists in arm and hand movements focusing on one joint at a time.

SUMMARY:
The purpose of this study is to develop an upper extremity robotic training system for use by people with stroke to practice arm and hand movement in the clinic.

DETAILED DESCRIPTION:
Each year in the U.S. over 400,000 people survive a stroke and approximately 80% of acute stroke survivors lose arm and hand movement skills. Movement impairments are typically treated with intensive, hands-on physical and occupational therapy for several weeks after the initial brain injury. Unfortunately, due to economic pressure on the U.S. health care system, stroke patients are receiving less therapy and going home sooner. Our goal for this study is to develop an upper extremity robotic training system for both acute and chronic stroke population to improve movement ability with intensive and repetitive movement in the clinic without continuous supervision from a therapist.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 73
* Sustained single stroke at least three months previously
* Minimal to moderate lost motor control of the arm after stroke

Exclusion Criteria:

* Concurrent severe medical problems
* Severe cognitive dysfunction
* Severe neglect or apraxia
* Severe visual deficits
* Significant subluxation of the shoulder
* Presence of severe elbow or wrist contracture
* Any metal implants or surgical clips or mechanical devices
* Metallic hardware on scalp region
* prior diagnosis of seizure and epilepsy
* severe migraine headache
* currently pregnant or lactating
* claustrophobic
* currently taking medication that lower seizure threshold

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Reinkensmeyer, Ph.D, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milot MH, Spencer SJ, Chan V, Allington JP, Klein J, Chou C, Bobrow JE, Cramer SC, Reinkensmeyer DJ. A crossover pilot study evaluating the functional outcomes of two different types of robotic movement training in chronic stroke survivors using the arm exoskeleton BONES. J Neuroeng Rehabil. 2013 Dec 19;10:112. doi: 10.1186/1743-0003-10-112. PMID 24354476

RESULTS

PARTICIPANT FLOW:
Groups:
- Individual Joints and Functional Multi-joints Tasks: Robotic group(Type I)
  Type II Robotic therapy (Individual joints only): Subjects participate in 11 weeks of training with the robotic device BONES, 3 days per week, 1 hour per day with a robot-assisted exercise program. The robotic exoskeleton assists in arm and hand movements as the patient play interactive computer games.
- Functional Multi-joints Activities and Individual Joints: Robotic group (Type II)
  Type I Robotic Group (Functional activities and individual joints): Subjects participate in 11 weeks of robotic training with the device: BONES (Biomimetic Orthosis Neurorehabilitation for Elbow and Shoulder) , 3 days per week, 1 hour per day with the robotic exercise program.
Period: Overall Study
Arm/Group | Individual Joints and Functional Multi-joints Tasks | Functional Multi-joints Activities and Individual Joints
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Type I Robotic Therapy (Functional Activities Then Individual Joint Exercises): Robotic group (Type I)
  Type I Robotic Group (Functional activities and individual joints): Subjects participate in 11 weeks of robotic training with the device: BONES (Biomimetic Orthosis Neurorehabilitation for Elbow and Shoulder), 3 days per week, 1 hour per day with the robotic exercise program involving multiple joints at the same time for the functional activities such as cleaning the window, driving a steering wheel, grocery shopping, etc; and then individual joint exercises focusing on one joint at a time with the individual joint exercises.
- Type II Robotic Therapy (Individual Joints Exercises Then Functional Activities): Robotic group (Type II)
  Type II Robotic therapy (Individual joints exercises then functional activities): Subjects participate in 11 weeks of training with the robotic device BONES, 3 days per week, 1 hour per day with a robot-assisted exercise program. The robotic exoskeleton assists in arm and hand movements as the patient perform individual joint exercises focusing on one joint at a time; and then functional activities like cleaning the window, driving a steering wheel, grocery shopping, etc for the functional activities.
- Total: Total of all reporting groups
Arm/Group | Type I Robotic Therapy (Functional Activities Then Individual Joint Exercises) | Type II Robotic Therapy (Individual Joints Exercises Then Functional Activities) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (7) | 60 (7) | 60 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Box & Blocks Test
Description: We measured the Box and Blocks Test scores at baseline evaluation, after each intervention, and at the 3-month follow up evaluation. Participants are instructed to move as many blocks as possible, one at a time, from one compartment in a box to a second compartment over a divider for a period of 60 seconds; each block that is moved is counted, and multiple blocks moved at the same time are counted as a single block. The higher scores indicate a better outcome.
Time Frame: Baseline, Post first intervention at 5 weeks, post second intervention at 11 weeks, and 3-month after the completion of the second intervention.
Measure: Mean (Standard Deviation); unit: blocks
Groups:
- Functional Multi-joint Training Then Individual Joint Training: Subjects participated in 4 weeks of training with the robotic device BONES, 3 days per week, 1 hour per day with a robot-assisted exercise program which focuses on functional multi-joint activities such as cleaning the windows, driving a steering wheel, grocery shopping, etc. Then, subjects performed individual joint exercises focusing on one joint at a time for another 4 weeks with 3 days per week and 1 hour per day with the robot-assisted exercise program.
- Individual Joint Training Then Functional Multi-joint Training: Subjects participated in 4 weeks of training with the robotic device BONES, 3 days per week, 1 hour per day with a robot-assisted exercise program which focuses on individual joint exercises, one joint at a time. Then, subjects performed the multi-joint functional training exercises for another 4 weeks with 3 days per week and 1 hour per day focusing on multi-joint activities such as cleaning the windows, driving a steering wheel, grocery shopping, etc.
Arm/Group | Functional Multi-joint Training Then Individual Joint Training | Individual Joint Training Then Functional Multi-joint Training
Number analyzed (Participants) | 10 | 10
blocks
  Baseline evaluation | 25 (11) | 36 (14)
  Post 1st Intervention | 29 (18) | 42 (14)
  Post 2nd Intervention | 31 (11) | 43 (13)
  3-month follow up evaluation | 28 (5) | 46 (9)

ADVERSE EVENTS:
Groups:
- Individual Joints: Robotic group(Type I)
  Type II Robotic therapy (Individual joints only): Subjects participate in 4 weeks of training with the robotic device BONES, 3 days per week, 1 hour per day with a robot-assisted exercise program. The robotic exoskeleton assists in arm and hand movements focusing on one joint at a time. Then, after one-week of a rest break, all subjects will return to participate in another 4 weeks of training with BONES again, 3 days per week with 1 hour per day, focusing on multi-joint activities such as cleaning the windows, driving a steering wheel, grocery shopping, etc.
- Functional Multi-Joint Activities: Robotic group (Type II)
  Type I Robotic Group (Functional Multi-joint activities): Subjects participate in 4 weeks of robotic training with the device: BONES (Biomimetic Orthosis Neurorehabilitation for Elbow and Shoulder), 3 days per week, 1 hour per day with the robotic exercise program focusing on multi-joint activities such as cleaning the windows, driving a steering wheel, grocery shopping, etc. Then, after a one-week rest break, all subjects will return to participate in another 4 weeks of training with BONES again, 3 days per week with 1 hour per day, focusing on individual joint exercises with one joint at a time.
Arm/Group | Individual Joints | Functional Multi-Joint Activities
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No